CLINICAL TRIAL: NCT04136431
Title: The Effects of Programmed Cryotherapy and Continuous Passive Motion in Patients After Computer-Assisted Total Knee Arthroplasty: A Prospective, Randomized Controlled Trial
Brief Title: Effects of Programmed Cryotherapy and Continuous Passive Motion After Computer-Assisted Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201102015B0
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2012-02

CONDITIONS: Patients With Osteoarthritis Undergoing CAS-TKA

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Programed cryotherapy and continuous passive motion
- Control group (Placebo Comparator)
  Interventions: Other: Unrogramed cryotherapy and continuous passive motion

INTERVENTIONS:
Other: Programed cryotherapy and continuous passive motion — The intervention group started to use a CPM machine and applied programed cryotherapy intermittently within one hour while returning to the ward on the day of surgery.
  Arms: Intervention group
Other: Unrogramed cryotherapy and continuous passive motion — A CPM machine and cryotherapy were not applied on the day of surgery while returning to the ward
  Arms: Control group

SUMMARY:
The hypothesis of this study was the patients, who received programed cryotherapy and CPM, had experienced less postoperative pain, joint swelling, and increased ROM following CAS-TKA.

DETAILED DESCRIPTION:
The International Association for the Study of Pain (IASP) has proposed the definition of pain as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage or described in terms of such damage. Therefore, adequate pain management and control of localized swelling and stiffness after TKA has become a priority because it is essential for improving patient satisfaction, prevention of complications, and enhancing quality of life by faster recovery. Systemic and local analgesics are the most common strategies for postoperative pain management in TKR. However, patients might experience nausea, vomiting, constipation, or respiratory failure due to opioid-related side effects, subsequently refusing to mobilize and delaying the rehabilitation program).

In addition to pain control, cryotherapy and continuous passive motion (CPM) are commonly used for TKA patients as non-pharmacological methods to reduce the postoperative pain and swelling and to increase the amount of knee flexion. The application of cryotherapy after TKA has been described extensively in the literature and is part of standard care globally. However, its benefits and value remain controversial due to the disparity in practice, such as differences in clinical protocols and the type of cryotherapy application. Continuous passive motion is a motorized device, which passively moves the knee joint within a certain range of motion (ROM) to decrease analgesics requirements, reduce the incidence of deep vein thrombosis, and increase ROM. But the effects of CPM remain contentious in the literature. Although controversial, cryotherapy and CPM have been used extensively as part of the standard postoperative management protocol for TKA patients without knowing its cost-effectiveness. However, the value of combined therapy of cryotherapy and CPM remains uncertainty and unclear following CAS-TKA.

The hypothesis of this study was the patients, who received programed cryotherapy and CPM, had experienced less postoperative pain, joint swelling, and increased ROM following CAS-TKA.

ELIGIBILITY:
Inclusion Criteria:

* primary and unilateral computer-assisted total knee arthroplasty

Exclusion Criteria:

* (1) patients who underwent bilateral TKAs, unicompartmental TKA or revision TKA
* (2) patients who had to remove previous implants or history of high-tibial or distal femoral corrective osteotomy
* (3) patients who were unable to response to the questionnaires.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03-07 (Actual); Primary Completion 2013-03-05 (Actual); Study Completion 2013-03-05 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Postoperative day 1
  Pain score. The scale is 0-10 where 0 is no pain and 10 is the worst pain
Numeric Rating Scale (NRS) | Postoperative day 4
  Pain score. The scale is 0-10 where 0 is no pain and 10 is the worst pain

SECONDARY OUTCOMES:
The short-form McGill Pain Questionnaire (SF-MPQ) | Postoperative day 1
  The SF-MPQ include 11 words of sensory subscale 4 words of affective subscale. These words are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe.
The short-form McGill Pain Questionnaire (SF-MPQ) | Postoperative day 4
  The SF-MPQ include 11 words of sensory subscale 4 words of affective subscale. These words are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe.
Thigh and calf circumference | Postoperative day 1
  The measurement of the thigh circumference was performed 15 cm proximal to the superior pole of the patella with a measurement tape, meanwhile 15 cm distal to the inferior pole of the patella for the calf circumference.
Thigh and calf circumference | Postoperative day 4
  The measurement of the thigh circumference was performed 15 cm proximal to the superior pole of the patella with a measurement tape, meanwhile 15 cm distal to the inferior pole of the patella for the calf circumference.
Range of motion of knee joints | Postoperative day 1
  A universal goniometer was used to measure extension and flexion arcs of the knee joints.
Range of motion of knee joints | Postoperative day 4
  A universal goniometer was used to measure extension and flexion arcs of the knee joints.

REFERENCES:
- [Derived] Chen MC, Lin CC, Ko JY, Kuo FC. The effects of immediate programmed cryotherapy and continuous passive motion in patients after computer-assisted total knee arthroplasty: a prospective, randomized controlled trial. J Orthop Surg Res. 2020 Sep 3;15(1):379. doi: 10.1186/s13018-020-01924-y. PMID 32883309